CLINICAL TRIAL: NCT00520351
Title: Comparison of Lens Care Regimens With a Silicone Hydrogel Lens (Emerald)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Craig Woods, Research Manager, CCLR
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P/265/07/L
Record Dates: First submitted 2007-08-21; First posted 2007-08-24 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: ClearCare
- 2 (Active Comparator)
  Interventions: Drug: Optifree Replenish

INTERVENTIONS:
Drug: ClearCare — contact lens care system
  Arms: 1
Drug: Optifree Replenish — contact lens care system
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate and compare, on a daily wear basis, the performance of two contact lens care solutions when used with silicone hydrogel soft contact lenses with regards to comfort and dryness symptoms.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate and compare, on a daily wear basis, the performance of two contact lens care solutions when used with silicone hydrogel soft contact lenses with regards to comfort and dryness symptoms by observing changes within the cornea and collecting subjective ratings

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 17 years of age and has full legal capacity to volunteer.
2. Has read, understood and signed an information consent letter.
3. Is willing and able to follow instructions and maintain the appointment schedule.
4. Is presently using either bi-weekly or monthly replacement lenses.
5. Has symptoms of ocular dryness as determined by specific pre-screening criteria.
6. Is correctable to a visual acuity of 6/9 or better (in each eye) with their habitual vision correction.
7. Has clear corneas and no active ocular disease.
8. Has had an ocular examination in the last two years.

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Is an asymptomatic lens wearer.
2. Is a daily disposable contact lens wearer.
3. Is a current extended wear contact lens wearer.
4. Currently uses one of the study lens care regimens.
5. Has any clinically significant blepharitis.
6. Has undergone corneal refractive surgery.
7. Is aphakic.
8. Has any active ocular disease.
9. Has any systemic disease affecting ocular health.
10. Is using any systemic or topical medications that may affect ocular health.
11. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
12. Is participating in any other type of clinical or research study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, M. Optom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, School of Optometry, University of Waterloo., Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study completion date is August 2008
Pre-assignment Details: Washout for 2 to 3 days following screening (wear spectacles only).
Groups:
- ClearCare First, Then Optifree Replenish: In Period 1, participants used ClearCare contact lens solution. There was a washout period of 2-3 days. Participants were then assigned to use OptifreeReplenish solution. In the first intervention participants were randomly assigned to use ClearCare first.
- Optifree Replenish First, Then ClearCare: In Period 1, participants used Optifree Replenish contact lens solution. There was a washout period of 2-3 days. Participants were then assigned to use ClearCare solution. In the first intervention, participants were randomly assigned to use Optifree Replenish first.
Period: First Intervention
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Started | 15 (Start date is Sep.06, 2007) | 15 (Start date is Sep.06, 2007)
Completed | 14 (End date is Feb.25, 2008) | 14 (End date is Feb.25, 2008)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (5.9) | 24.1 (4.4) | 24.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Visual Acuity
Description: High Contrast Visual Acuity with contact lenses, was measured using standardized and computer generated logMAR chart.
  10 Sloan letters adopted. VA chart's target size varied from logMAR 1.0 to -0.40 in 0.1 logMAR step.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Number analyzed (Participants) | 28 | 28
logMAR | -0.04 (0.06) | -0.04 (0.06)

2. Primary Outcome: Low Contrast Visual Acuity
Description: Low Contrast Visual Acuity with contact lenses, was measured using standardized and computer generated logMAR chart.
  10 Sloan letters adopted. VA chart's target size varied from logMAR 1.0 to -0.40 in 0.1 logMAR step.
Time Frame: 2 weeks
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Number analyzed (Participants) | 28 | 28
logMAR | 0.26 (0.07) | 0.25 (0.08)

3. Primary Outcome: In-vivo Wettability
Description: Pre-lens non-invasive tear breakup time
Time Frame: 2 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Number analyzed (Participants) | 28 | 28
Seconds | 7.06 [5.8 to 8.3] | 6.54 [5.7 to 7.4]

4. Primary Outcome: Subjective Comfort Rating
Description: Numeric rating scale was administered. Comfort ratings (0 - 100), 0 = Very poor comfort and 100 = Excellent comfort.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Number analyzed (Participants) | 28 | 28
Units on a scale | 82.5 [70.3 to 94.8] | 81.3 [64.9 to 97.8]

ADVERSE EVENTS:
Time Frame: 6 months
Description: An adverse event included any undesirable clinical occurrence in a participant, whether it was considered to be device-related or not.
Arm/Group | ClearCare First, Then Optifree Replenish | Optifree Replenish First, Then ClearCare
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days